CLINICAL TRIAL: NCT01971996
Title: Measuring the Cerebral Oxygen Saturation With NIRS Sensor Placed on the Forehead of Patients in the Prone Position. How Does the External Pressure Affect the Measurement.
Brief Title: Measuring the Effect of External Pressure on the Regional Cerebral Oxygen Saturation Monitored by Near-infrared Spectroscopy(NIRS) Technology
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Johnny Andersen, M.D., Glostrup University Hospital, Copenhagen
Other Study IDs: H-4-2013-FSP
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Anaesthesia
Keywords: Near infrared Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lumbar spine surgical patients: Patients undergoing lumbar spine surgery in the prone position

SUMMARY:
During general anaesthesia, to ensure sufficient oxygen supply to the brain, the NIRS technology can be used. It consist of two sensors placed on the forehead, and measures the oxygen saturation of the tissue underneath the sensor. For patients undergoing back surgery placed in the prone position, the NIRS measurement will be affected, because the weight of the head will produce a pressure on the sensors. We wish to investigate how much the measurement is affected. Furthermore we plan to lift the head to remove the pressure, and record the time needed for the measurements to return to baseline.

DETAILED DESCRIPTION:
When placed in the prone position an external pressure is applied to the NIRS sensor. This pressure changes the amount of blood in the underlying tissue and thereby has an influence on the regional cerebral oxygen saturation measured. We wish to investigate to which extend this value is affected by the external pressure. Furthermore by lifting the head we want to investigate how long takes for the measurements to return to baseline (no pressure in the supine position).

Patients will receive written and oral information about the study, when seen by an anaesthesiologist prior to surgery. Before the anaesthesia one NIRS sensors is placed on the right side of the forehead, avoiding til frontal sinus, and one NIRA sensor is placed on the left musculus deltoideus. The patient is placed in the prone position with the head in af prone-view face mask. Measurements will start after 30 minutes with no change in infusion rate of anaesthetic and no inotropics administered. Registration of NIRS measurements will be done every 15 seconds, first five minutes without intervention, then five minutes with headlift, and last five minutes without interventions. Blood pressure, pulse, saturation, end-tidal carbon dioxide and temperature, will be recorded. Registration wil be om case report forms.

ELIGIBILITY:
Inclusion Criteria:

* Surgery in the lumbar spine, in the prone position, with the head in a proneview facemask
* Free and painless movement of the neck

Exclusion Criteria:

* Known cervical spine pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lumbar spine surgury, and are placed in the prone position
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in the regional cerebral oxygen saturation | 15 seconds
  Measured by Near Infrared Spectroscopy

SECONDARY OUTCOMES:
The duration before the steady state in the regional cerebral oxygen saturation is obtained after changing the head position. | 15 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Johnny DH Andersen, M.D., Principal Investigator — University of Copenhagen, Glostrup Hospital, Denmark; Hanna Siegel, M.D., Principal Investigator — University of Copenhagen, Glostrup Hospital, Denmark
Locations (1):
- University of Copenhagen, Glostrup Hospital, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Derived] Siegel H, Andersen JD, Nielsen RV, Lorentzen K, Olsen KS. Measuring regional cerebral oxygen saturation during surgery in the prone position. Eur J Anaesthesiol. 2016 Feb;33(2):154-5. doi: 10.1097/EJA.0000000000000289. No abstract available. PMID 26086290